CLINICAL TRIAL: NCT04598217
Title: The Effect of Virtual Reality on Preoperative Anxiety in Septorhinoplasty Patients
Brief Title: Is Virtual Reality a Non-pharmacological Premedication?
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Çağdaş Baytar, assistant professor, Zonguldak Bulent Ecevit University
Other Study IDs: 2020/19
Record Dates: First submitted 2020-10-06; First posted 2020-10-22 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Anxiety
Keywords: Virtual Reality; Anxiety; Premedication
MeSH Terms: conditions — Anxiety Disorders | interventions — Anesthesiologists

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: anesthesiologist — non-interventional observational

SUMMARY:
Preoperative anxiety of patients who will undergo septorhinoplasty surgery will be measured and their hemodynamic parameters will be recorded afterwards. Then, a video will be shown to the patients through virtual reality glasses and the effect of this application on their anxiety will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II risk group
* Will be operated under general anesthesia under elective conditions
* Going to undergo surgery for septoplasty / rhinoplasty
* Patients whose informed consent was read and approved

Exclusion Criteria:

* Those who do not want to participate in the study
* ASA III - IV-V patients
* Psychiatric-Cognitive dysfunction
* Claustrophobia
* Patients using sedative and narcotic drugs
* Alcohol-drug addicts
* Blind or deaf patients
* Patients who cannot speak Turkish

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65 who will undergo septorhinoplasty surgery
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
to reduce preoperative anxiety | through study completion, an average of 3 months
  Investigation of the effect of virtual reality applications on preoperative anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No